CLINICAL TRIAL: NCT07172191
Title: Manipulation of the Enteral Microbiome by Fecal Microbiota Transplantation Among Adult Patients With Malignant Hematological Diseases
Brief Title: Fecal Microbiota Transplantation Among Adult Patients With Hematological Malignancies
Acronym: HEMAT-FMT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Del-Pest Central Hospital - National Institute of Hematology and Infectious Diseases (Other)
Responsible Party: Principal Investigator, Bálint Gergely Szabó, M.D. Ph.D., Del-Pest Central Hospital - National Institute of Hematology and Infectious Diseases
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMAT-FMT; 15754-3/2023/EÜIG (Other: Scientific and Research Ethics Committee of the Hungarian National Medical Scientific Council)
Record Dates: First submitted 2025-08-25; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Malignant Hematologic Neoplasm
Keywords: Malignant hematologic neoplasm; Fecal microbiota transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients for inclusion are stratified into different interventional subgroups based on four differenc clinical indications for FMT as intervention:
  1. patient group: elimination of documented MDR colonization,
  2. patient group: treatment of active C. difficile infection,
  3. patient group: enteral microbiome restoration following autologous and allogeneic hematopoietic stem cell transplantation,
  4. patient group: treatment of corticosteroid-refractory acute gastrointestinal GvHD (see later).
  Control groups not receiving FMT as intervention are selected either: 1) from patients who possess the same clinical severity/stage and clinical indication for FMT, but do not agree to participate in the study or not eligible for technical reasons, or 2) randomly selected from patients without malignant hematological diseases and are hospitalized at our center. Patient recruitment is conducted consecutively, and a 1:2 ratio for case-control matching is followed during inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Experimental): Patients receiving fecal microbiota transplantation (FMT) for different clinical reasons
  Interventions: Biological: Fecal Microbial Transplantation
- non-FMT (No Intervention): Patients not receiving fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — The technical implementation of FMT procedure is consistent with the methodological letter issued by the National Public Health Center of Hungary. FMT is performed via nasogastric tube with suspended fresh stool graft obtained from a pre-selected stool donor. Following FMT, the patient is observed for 24 hours at our center. The process is supervised and performed by the lead researcher.
  Arms: FMT

SUMMARY:
In Hungary - in comparison to other member states of the European Union - about 75000 new cases of cancer are diagnosed annually, from which approximately 4500-5000 patients suffer from so-called malignant hematological diseases. This disease group includes various leukemias (blood cancers) and lymphomas (lymph node cancers). Chemotherapy for patients with malignant hematological diseases is particularly difficult to bear, as it affects the entire body, including the "good" gut bacteria living inside, and recovery can take several years. Due to the decrease of the "good" gut bacteria during treatment, patients are more prone to acquiring various difficult-to-treat infections, which can lead to deterioration of quality of life, prolonged hospitalization, and in the worst cases, death. The method outlined in this research plan is called fecal microbiota transplantation, during which stool from a healthy person is introduced into the body of the sick patient. The "good" gut bacteria present in the stool then restore the patient's entire gut flora (the process is somewhat similar to the use of probiotics available on the market, but it is a much more effective method). This research aims to assess the success of fecal microbiota transplantation in adults with malignant hematological diseases over a long-term follow-up period, thus contributing to the restoration of their acceptable quality of life.

DETAILED DESCRIPTION:
Fecal microbiota transplantation (FMT) is currently a widely accepted method of manipulating enteric microbiome, and is an internationally recommended procedure in the treatment for Clostridioides (formerly Clostridium) difficile (C. difficile) infection. The goal of FMT is to restore physiological gut microbiome through natural competition, by administering a stool graft harvested from a healthy person. FMT not only eliminates C. difficile-induced colitis, but also colonization of multidrug-resistant bacterial/fungal species, and certain types of intestinal epithelial damage occuring in some medical conditions. In recent years due to pleiotropic effects of FMT, scientific interest has turned towards adult patients with malignant hematological diseases, since all of the pathological conditions mentioned earlier occur during clinical care in this population, due to detrimental effects of immuno-chemotherapy. Based on promising preliminary results, FMT could be a successful, easily implementable intervention for these patients in the future.

Therefore, the aim of this study is to perform FMTs in four indication groups among adult patients with malignant hematological diseases treated at South Pest Central Hospital - National Institute of Hematology and Infectious Diseases (Budapest, Hungary), followed by a 180-day follow-up period, during which standardized clinical, laboratory, imaging, and microbiological data are collected. In addition, a high-resolution microbiome analys to monitor microbiological changes of recipient pre-/post-FMT blood and stool samples is planned, in collaboration with Departmental Group of Infectious Diseases and Institute of Medical Microbiology of Semmelweis University (Budapest, Hungary).

This study aims to assess both the bacterial and fungal components of the enteric microbiome in adult patients receiving routine clinical care for malignant hematological diseases, and to explore the potential of manipulating the microbiome through fecal microbiota transplantation (FMT). The hypothesis is that microbiome manipulation with FMT in these patients may induce a successful and sustained response by restoring the physiological intestinal microbiome, a premise that this long-term, comprehensive clinical and microbiological follow-up study seeks to support.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (diagnosis age ≥18 years) with malignant hematological disease treated at our center, and
2. Capable of giving written informed consent after decision-making, and
3. Documented patient colonization with MDR bacterial or fungal isolates, or
4. Active C. difficile infection, or
5. Patient has undergone autologous or allogeneic hematopoietic stem cell transplantation, or
6. Ongoing corticosteroid-refractory acute gastrointestinal GvHD.

Exclusion criteria (one or more must be met):

1. Active bacterial or fungal bloodstream infection requiring antimicrobial therapy, or
2. Peripheral blood absolute neutrophil count <0.5 G/l on ≥7 consecutive days before planned FMT with maximum dose of administered G-CSF, or
3. Pressor-refractory septic shock, or
4. Major gastrointestinal bleeding within 7 consecutive days before planned FMT, or
5. Any pathological process inhibiting successful or safe nasogastric tube insertion, or
6. Lack of written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease activity | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Disease activity: hematological remission vs. relapse, GvHD activity. Disease activity of the malignant hematological underlying disease (hematological remission vs. relapse) is defined according to the published methodological recommendations by the National Comprehensive Cancer Network and the European Hematology Association (or the American Society of Hematology, if neither has specific guidance), specifically for each disease. GvHD activity is defined according to the published methodological recommendations of the European Bone Marrow Transplantation Society.

SECONDARY OUTCOMES:
Reducibility of applied immunosuppressive pharmacotherapy | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Reducibility of applied immunosuppressive pharmacotherapy. The reducibility of immunosuppressive and antimicrobial pharmacotherapy is determined based on the number of active substances and changes in dose intensity.
Reducibility of applied antimicrobial pharmacotherapy | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Reducibility of applied antimicrobial pharmacotherapy. The reducibility of immunosuppressive and antimicrobial pharmacotherapy is determined based on the number of active substances and changes in dose intensity.
Survival | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared controls
  Survival: total and progression-free survival. Total survival: the patient does not die during the follow-up period. Progression-free survival: during the follow-up period, the stage of the malignant hematological underlying disease documented at enrollment does not change or improves (partial or complete hematological remission occurs), and the patient does not die. The activity of the malignant hematological underlying disease is defined according to the published methodological recommendations by the National Comprehensive Cancer Network and the European Hematology Association (or the American Society of Hematology, if neither has specific guidance), specifically for each disease.
Clinical cure of C. difficile infection | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Clinical cure of C. difficile infection: we apply the guidelines of the European Society of Clinical Microbiology and Infectious Diseases to define clinical cure

OTHER OUTCOMES:
Loss of colonization with multidrug-resistant bacterial or fungal isolates | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Loss of colonization with multidrug-resistant bacterial or fungal isolates: Colonization cannot be confirmed by standard microbiological culturing from samples taken from investigated anatomical locations (see earlier). The definitions of multidrug resistance are based on the recommendations of Magiorakos et al. (Clinical Microbiology and Infection, 2012) and Kristóf et al. (Mikrobiológiai Körlevél, 2021 [in Hungarian]).
Loss of C. difficile colonization | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Loss of C. difficile colonization: The presence of C. difficile GDH antigen and "A+B" toxins cannot be confirmed in the regularly stored and transported stool sample of an asymptomatic person. We apply the guidelines of Debast et al. (Clinical Microbiology and Infection, 2014) for detection.
Regeneration of blood and gut microbiome after autologous and allogeneic stem cell transplantation | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Regeneration of blood and gut microbiome after autologous and allogeneic stem cell transplantation: Based on abundance analysis performed by 16S metagenome sequencing of collected blood and stool samples.
Regeneration of blood and gut microbiome during GvHD | On Day 7, Day 30, Day 60 and Day 180, since the intervention, compared to baseline and controls
  Regeneration of blood and gut microbiome during GvHD: Based on abundance analysis performed by 16S metagenome sequencing of collected blood and stool samples.

CONTACTS AND LOCATIONS:
Locations (1):
- South Pest Central Hospital, National Institute of Hematology and Infectious Diseases, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author upon reasonable request. Restrictions apply to the availability of raw patient-level data due to ethical and privacy considerations.

REFERENCES:
- [Background] Deeg HJ. How I treat refractory acute GVHD. Blood. 2007 May 15;109(10):4119-26. doi: 10.1182/blood-2006-12-041889. Epub 2007 Jan 18. PMID 17234737
- [Background] Pession A, Zama D, Muratore E, Leardini D, Gori D, Guaraldi F, Prete A, Turroni S, Brigidi P, Masetti R. Fecal Microbiota Transplantation in Allogeneic Hematopoietic Stem Cell Transplantation Recipients: A Systematic Review. J Pers Med. 2021 Feb 4;11(2):100. doi: 10.3390/jpm11020100. PMID 33557125
- [Background] Kaito S, Toya T, Yoshifuji K, Kurosawa S, Inamoto K, Takeshita K, Suda W, Kakihana K, Honda K, Hattori M, Ohashi K. Fecal microbiota transplantation with frozen capsules for a patient with refractory acute gut graft-versus-host disease. Blood Adv. 2018 Nov 27;2(22):3097-3101. doi: 10.1182/bloodadvances.2018024968. PMID 30446486
- [Background] DeFilipp Z, Peled JU, Li S, Mahabamunuge J, Dagher Z, Slingerland AE, Del Rio C, Valles B, Kempner ME, Smith M, Brown J, Dey BR, El-Jawahri A, McAfee SL, Spitzer TR, Ballen KK, Sung AD, Dalton TE, Messina JA, Dettmer K, Liebisch G, Oefner P, Taur Y, Pamer EG, Holler E, Mansour MK, van den Brink MRM, Hohmann E, Jenq RR, Chen YB. Third-party fecal microbiota transplantation following allo-HCT reconstitutes microbiome diversity. Blood Adv. 2018 Apr 10;2(7):745-753. doi: 10.1182/bloodadvances.2018017731. PMID 29592876
- [Background] Biernat MM, Urbaniak-Kujda D, Dybko J, Kapelko-Slowik K, Prajs I, Wrobel T. Fecal microbiota transplantation in the treatment of intestinal steroid-resistant graft-versus-host disease: two case reports and a review of the literature. J Int Med Res. 2020 Jun;48(6):300060520925693. doi: 10.1177/0300060520925693. PMID 32527171
- [Background] Battipaglia G, Malard F, Rubio MT, Ruggeri A, Mamez AC, Brissot E, Giannotti F, Dulery R, Joly AC, Baylatry MT, Kossmann MJ, Tankovic J, Beaugerie L, Sokol H, Mohty M. Fecal microbiota transplantation before or after allogeneic hematopoietic transplantation in patients with hematologic malignancies carrying multidrug-resistance bacteria. Haematologica. 2019 Aug;104(8):1682-1688. doi: 10.3324/haematol.2018.198549. Epub 2019 Feb 7. PMID 30733264
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):e1-e48. doi: 10.1093/cid/cix1085. PMID 29462280
- [Background] Debast SB, Bauer MP, Kuijper EJ; European Society of Clinical Microbiology and Infectious Diseases. European Society of Clinical Microbiology and Infectious Diseases: update of the treatment guidance document for Clostridium difficile infection. Clin Microbiol Infect. 2014 Mar;20 Suppl 2:1-26. doi: 10.1111/1469-0691.12418. PMID 24118601